CLINICAL TRIAL: NCT07094425
Title: Intensive Care Unit-acquired Heart Failure in Critically Ill: the ICU-HF Study
Acronym: ICU-HF
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan J Schaller, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ICU-HF
Record Dates: First submitted 2025-07-18; First posted 2025-07-30 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; ICUAW
Keywords: Critical Illness
MeSH Terms: conditions — Heart Failure; Critical Illness | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically Ill Patients: Patients admitted to Intensive Care Unit
  Interventions: Diagnostic Test: transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: transthoracic echocardiography — Transthoracic echocardiography (TTE) is a non-invasive method for assessing cardiac morphology and function. As part of the study protocol, TTE will be performed at the time of study inclusion (within the first 24 hours after ICU admission), on day 3, day 7, and day 14, followed by weekly assessments (until discharge from the ICU), as well as on the day of planned ICU or hospital discharge.
  To verify skeletal muscle mass in relation to myocardial mass and its changes over the course of the ICU stay, bioelectrical impedance analysis (BIA) will be performed at the time points mentioned above.
  Other Names: body impedance analysis

SUMMARY:
Critically ill patients in intensive care units (ICUs) are exposed to a wide range of complications that can affect long-term morbidity and mortality. Not only the initial diagnosis at the time of admission may lead to complications; the ICU stay itself can also be associated with specific disease patterns.

One of the most frequent complications of intensive care treatment is the loss of skeletal muscle mass. Muscle atrophy can be detected in up to 17% of all critically ill ICU patients. This is accompanied by a neuromuscular organ dysfunction collectively referred to as Intensive Care Unit Acquired Weakness (ICUAW). Milder forms of ICUAW are present in up to 40% of all ICU patients, which corresponds to approximately 1.2 million individuals per year in Germany alone. These patients face a multitude of long-term complications and have an increased mortality risk that may persist for up to five years after ICU discharge.

To date, the definition of ICUAW is limited to the skeletal musculature of critically ill patients. It remains unclear whether an ICU stay also affects other muscle groups, such as the myocardium. A first retrospective study demonstrated a significant reduction in cardiac muscle mass in critically ill ICU patients. However, the clinical implications of this loss of myocardial mass and the contributing factors remain uncertain. In addition, the patient cohort was highly heterogeneous regarding the initial diagnosis, the intensive care therapies performed (e.g., invasive ventilation), and the findings were based on a small sample size of just 44 patients.

Another study investigated the association between skeletal muscle atrophy and myocardial structure in a cohort of 378 community-dwelling older adults. They showed that a decrease in skeletal muscle mass was also accompanied by a reduction in myocardial mass. Furthermore, they found a correlation between skeletal muscle atrophy and reductions in left ventricular and left atrial dimensions. However, it remains unclear whether a reduction in myocardial mass is associated with heart failure.

Heart failure is associated with a significantly increased risk of long-term morbidity and mortality. The diagnosis and staging of heart failure is primarily based on morphological assessment via transthoracic echocardiography (TTE), in combination with laboratory biomarkers (e.g., NT-proBNP), and the patient's subjective functional impairment as classified by the New York Heart Association (NYHA). Identifying heart failure is clinically relevant, as optimized pharmacologic therapy can lead to significant improvements in cardiac function and positively impact long-term survival.

The aim of this study is to investigate the impact of intensive care treatment on myocardial mass and to assess a potential correlation with heart failure. Measurement of myocardial mass and evaluation of heart failure will be performed via transthoracic echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients aged ≥ 18 years
* Initiation of mechanical ventilation within the first 24 hours after ICU admission
* Expected duration of ICU stay of at least 3 days

Exclusion Criteria:

* Language barriers
* Expected death during ICU stay or planned transition to best supportive care
* Known allergy to electrode gel
* Ultrasound not technically feasible (e.g., due to extensive wounds, skin rash, or dressings)
* Patients with a pacemaker or similar electronic devices for whom bioelectrical impedance analysis (BIA) is contraindicated
* Patients with severe aortic valve stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes critically ill adults aged ≥18 years who require mechanical ventilation started within 24 hours of ICU admission and are expected to stay in the ICU for at least 3 days.
  Exclusion criteria are: language barriers preventing informed consent or participation; expected death during ICU stay or planned shift to best supportive care; allergy to electrode gel; inability to perform transthoracic ultrasound or bioimpedance analysis due to extensive wounds, skin conditions, or dressings; presence of implantable electronic devices (e.g., pacemakers) contraindicating bioimpedance measurement; and severe aortic valve stenosis confirmed clinically or by prior echocardiography.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of myocardial mass during the course of intensive care in critically ill patients, assessed by transthoracic echocardiography according to ASE/EACVI guidelines based on left ventricular wall thickness and diameter measurements. | Within 14 days

SECONDARY OUTCOMES:
Correlation between the reduction of myocardial mass (assessed by transthoracic echocardiography) and the occurrence or progression of systolic heart failure (based on echocardiographic left ventricular ejection fraction measurements) | Within 14 days
Correlation between the reduction of myocardial mass (assessed by transthoracic echocardiography) and the occurrence or progression of diastolic heart failure (based on echocardiographic left ventricular ejection fraction measurements) | Within 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Medical University of Vienna, Vienna, Vienna, Austria
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No